CLINICAL TRIAL: NCT06543212
Title: Eye Alignment and Eye Control Changes Through Follow up Period After Application of Eye Exercises Post Strabismus Surgery
Status: Completed | Type: Observational
Sponsor: Amany Refaat Mohamed Abdel Wahid (Other)
Responsible Party: Sponsor-Investigator, Amany Refaat Mohamed Abdel Wahid, lecturer at faculty of physical therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/004678
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Strabismus; Intermittent
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group continues with physiotherapy: Group continues with physiotherapy training in follow up period after last session of physiotherapy program post strabismus surgery.
  Interventions: Other: physiotherapy exercises
- group doesn't continue with physiotherapy: Group doesn't continue with physiotherapy training in follow up period after last session of physiotherapy program post strabismus surgery

INTERVENTIONS:
Other: physiotherapy exercises — physiotherapy exercises to improve eye alignment and eye control post strabismus surgery
  Groups: group continues with physiotherapy

SUMMARY:
The aim of this study is to determine the patient status through its follow up period and weather the eye alignment and eye control are as the same as the last physiotherapy treatment session or there is any deterioration of them.

DETAILED DESCRIPTION:
This study is quantitative cohort observational study. The study depends on following a group of participants over a period of time ( 2 months after completed physiotherapy training program for 3 months to improve eye alignment and eye control post strabismus surgery ).

Through the study, there is observation to the changes in certain quantitative variables ( eye alignment and eye control ).

ELIGIBILITY:
Inclusion Criteria:

* Patients are both males and females.
* Their age will range from (5-15) years.
* All Patients received physiotherapy training for improving eye alignment and eye control.
* Patients applied the physiotherapy rehabilitation program for 3 months with the physiotherapist.
* All Patients complete their physiotherapy training sessions for improving eye alignment and eye control
* All Patients have a history of strabismus surgery.
* Intermittent exotropia was the type of strabismus which included to the study.

Exclusion Criteria:

* - Patient who didn't receive physiotherapy training program for improving eye control and eye alignment post strabismus surgery.
* Patient who didn't complete the physiotherapy training program for 3 months.
* Muscular disorders that will impair performance during training.
* Any organic lesion in the eye.
* Neurological disorders.
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population from both groups will be selected from Research Institute of Ophthalmology and completed physiotherapy training program for 3 months to improve eye alignment and eye control post strabismus surgery.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Eye deviation by prism-cover test | 3 months
  This test is used to quantify the movement of deviating eye
Measurement of eye control by Intermittent Exotropia Control Scale | 3 months
  The level of control will be evaluated in each patient at both distance and near fixation using Intermittent Exotropia Control Scale. The scale ranges from 0 (phoria, best control) to 5 (constant exotropia, worst control).

CONTACTS AND LOCATIONS:
Overall Officials: Amany Abdel Wahid, Post doctor, Study Director — Lecturer at faculty of physical therapy, Cairo University
Locations (1):
- Cairo University, Giza, Giza Governorate, Egypt